CLINICAL TRIAL: NCT01037660
Title: Effects of Lipemia and Metformin on Endothelial Function
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Principal Investigator, Naomi M Hamburg, PI, Boston University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-23660
Record Dates: First submitted 2009-12-19; First posted 2009-12-23 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Cardiovascular Disease
Keywords: endothelium; cardiovascular disease; dietary fat; insulin resistance
MeSH Terms: conditions — Cardiovascular Diseases; Insulin Resistance | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Metformin (Experimental): Metformin
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin 1 gram per day

SUMMARY:
Eating a diet high in fat contributes to the development of atherosclerosis (hardening of the arteries). Acute fat consumption increases levels of fat in the blood and temporarily reduces the ability of blood vessel to dilate (open up to carry additional blood). A similar response is observed during infusion of Intra-Lipid (a fat emulsion used for intravenous nutrition). The present study is designed to help us understand the effects of a fat load on blood vessel function. We will measure arterial dilation using non-invasive techniques before and at the end of a 5-hour infusion of Intra-Lipid in healthy subjects. Subjects will then take the approved drug metformin for two weeks and return for repeat studies of endothelial function with Intra-Lipid infusion. We expect that metformin will help preserve the normal function of blood vessels during a fat load. This study will help us understand how fat affects blood vessels and therefore will advance our knowledge of the development of atherosclerosis and potentially lead to improved methods to prevent and treat heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Pregnancy (defined as positive urine pregnancy test)
* Diabetes Mellitus (Clinical history or random blood glucose>140 mg/dl)
* Hypertension (Clinical history or SBP>140 or DBP>90 mmHg)
* History of adverse reaction to metformin
* Abnormal renal function (Serum creatinine>1.4 mg/dl)
* Abnormal liver function (AST or ALT greater than two times the upper limit of normal)
* Administration of iodinated contrast within 7 days
* History of congestive heart failure
* Abnormal clotting parameters (INR>1.5 or PTT>40 sec)
* Anemia (HCT<30%)
* Allergy to soy or egg
* Allergy to heparin
* The potential subject plans to perform heavy exercise in the setting of low calorie intake during the period of the study such as running or competitive road or bicycle racing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2005-09 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Brachial artery flow-mediated dilation | 6 hours

SECONDARY OUTCOMES:
blood lipid levels | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Hamburg, MD, Principal Investigator — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No